CLINICAL TRIAL: NCT06666699
Title: Design Optimization of RIVOS EUS Access Device - A Feasibility Study
Brief Title: RIVOS Feasibility (MBO)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been withdrawn per decision of Sponsor.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: E7189
Record Dates: First submitted 2024-10-11; First posted 2024-10-31 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Malignant Biliary Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- RIVOS (Experimental)
  Interventions: Device: EUS access device

INTERVENTIONS:
Device: EUS access device — The intervention involves the use of an EUS access device to gain access to the bile duct via hepaticogastrostomy.

SUMMARY:
The goal of this clinical trial is to assess basic feasibility, safety, and performance of an EUS access device in patients with malignant biliary obstruction who are indicated to receive EUS-guided hepaticogastrostomy for biliary drainage. The main questions it aims to answer are:

* Can the device be used to gain and maintain access to target anatomy?
* Does the device have a clinically acceptable safety profile?
* How does the device perform overall?

All patients will undergo a hepaticogastrostomy procedure and be followed for 7 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with malignant biliary obstruction and who is indicated to receive EUS-guided hepaticogastrostomy for biliary drainage, as documented by dilated left hepatic duct and hyperbilirubinemia
* Patient who failed ERCP (e.g., inability to access the obstructed biliary system via a transpapillary route) or for whom ERCP is not an option (e.g., due to altered anatomy, gastric outlet obstruction)
* 18 years of age or older
* Patient willing and able to provide written informed consent and comply with specified study visits

Exclusion Criteria:

* Patient whose general medical condition and degree of respiratory failure would not allow them to tolerate endoscopy and/or the manipulation required to perform the study procedure
* Abnormal coagulopathy:

  * INR >1.5 and not correctable
  * presence of bleeding disorder
  * platelets <50,000 mm3
* Patient with contraindication to use of electrical devices
* Female of childbearing potential with a positive pregnancy test prior to the procedure or who intends to become pregnant during the study
* Patient from a vulnerable population
* Current participation in another investigational drug or device study that could interfere with the endpoints of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Day 0 Study Procedure
  Defined as (1) access of the target biliary duct, as confirmed via imaging, (2) ability to advance a wire to guide the procedure through the access cannula after the sharp is removed, and (3) ability to create a cautery fistula for accessory device passage
Safety | Day 0 Study Procedure through Day 7 Post-Study Procedure
  Study device- and study procedure-related serious adverse events
Device Performance | Day 0 Study Procedure
  Evaluated per the following criteria (1) ability to gain access to the target structure, (2) ability to maintain access to the target structure, (3) ability to visualize device during necessary procedural steps, and (4) ability to create a cautery fistula for accessory device passage

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Lakhtakia, MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (3):
- Ghent University Hospital, Ghent, Belgium
- Georges Pompidou European Hospital, Paris, France
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No